CLINICAL TRIAL: NCT04486430
Title: A Phase II, Double-blind, Randomized, Placebo-controlled, Multi-center Study to Assess the Efficacy and Safety of the Salfaprodil for Injection in Patients With Acute Ischemic Stroke
Brief Title: Efficacy and Safety Study of Neu2000KWL for Acute Ischemic Stroke Patients Within 6 Hours of Onset
Acronym: Salfaprodil
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Zhejiang Apeloa Jiayuan Pharmaceutical Co. Ltd. (Unknown); Subei People's Hospital of Jiangsu Province (Other); The First Hospital of Jilin University (Other); First Hospital of China Medical University (Other); General Hospital of Shenyang Military Region (Other); The First Affiliated Hospital of BaoTou Medical College (Other); Xuanwu Hospital, Beijing (Other); Peking University First Hospital (Other); Peking University Third Hospital (Other); Tianjin First Central Hospital (Other); Tianjin Huanhu Hospital (Other); Hebei Medical University Third Hospital (Other); The Second Hospital of Hebei Medical University (Other); Hebei General Hospital (Other); Second Hospital of Shanxi Medical University (Other); Shandong Provincial Hospital (Other Government); Qilu Hospital of Shandong University (Other); The First Affiliated Hospital of Soochow University (Other); Nanjing PLA General Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Minhang Central Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Xiangya Hospital of Central South University (Other); Guangzhou First People's Hospital (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Nanfang Hospital, Southern Medical University (Other); First Affiliated Hospital of Jinan University (Other); Tongji Hospital (Other); The Central Hospital of Lishui City (Other); Shanghai Pudong New Area People's Hospital (Other); Inner Mongolia Baogang Hospital (Other); Daqing Oil Field Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Vice President of Tian Tan Hospital, Director of Neurology Center, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YWZC-PLJY0125
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2017-01

CONDITIONS: Stroke; Cerebral Infarction
Keywords: Stroke; the Salfaprodil for injection; Neu2000KWL; Neuroprotection; glutamate; free radical
MeSH Terms: conditions — Stroke; Cerebral Infarction | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Neu2000KWL 2750mg dose group (Experimental): Low dose group
  Interventions: Drug: Neu2000KWL
- Neu2000KWL 5250mg dose group (Experimental): Middle dose group
  Interventions: Drug: Neu2000KWL
- Neu2000KWL 6000mg dose group (Experimental): High dose group
  Interventions: Drug: Neu2000KWL
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Neu2000KWL — 1st infusion of 500mg in patients within 6 hours following ischemic stroke onset followed by 9 consecutive infusions of 250 mg at intervals of 12 hours
  Other Names: Salfaprodil for injection
  Arms: Neu2000KWL 2750mg dose group
Drug: Neu2000KWL — 1st infusion of 750mg in patients within 6 hours following ischemic stroke onset followed by 9 consecutive infusions of 500 mg at intervals of 12 hours
  Other Names: Salfaprodil for injection
  Arms: Neu2000KWL 5250mg dose group
Drug: Neu2000KWL — 1st infusion of 1500mg in patients within 6 hours following ischemic stroke onset followed by 9 consecutive infusions of 500 mg at intervals of 12 hours
  Other Names: Salfaprodil for injection
  Arms: Neu2000KWL 6000mg dose group
Drug: Placebos — 1st infusion of the same volume of saline in patients within 6 hours following ischemic stroke onset followed by 9 consecutive infusions of the same volume of saline at intervals of 12 hours
  Arms: Placebo

SUMMARY:
The purpose of the study is to explore safety and efficacy of Salfaprodil administration for patients with acute ischemic stroke within 6 hours of onset.

DETAILED DESCRIPTION:
The present study is to investigate safety and efficacy of Neu2000, a multi-target neuroprotectant acting as a moderate NR2B-selective NMDA receptor antagonist and potent antioxidant, in acute ischemic stroke patients within 6 hours of onset. Compared to NMDA antagonists or antioxidants, improved efficacy and therapeutic time window of Neu2000 have been well documented in four animal models of stroke. Notable Safety of Neu2000 has been demonstrated in 168 human subjects conducted in the US and China as well as animals.

In the present phase II study, patients with acute ischemic stroke within 6 hours of onset would be assigned randomly to one of four groups as follows:

* Group A receiving 2.75g Neu2000KWL for 5 days
* Group B receiving 5.25g Neu2000KWL for 5 days
* Group C receiving 6.00g Neu2000KWL for 5 days
* Group D receiving placebo for 5 days

Patients will receive intravenous infusion of the clinical study drug twice a day at 12±1 hour intervals for 5 days.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged between 35 and 75 years;
2. acute ischemic stroke patients in internal carotid artery system within 6 hours of onset;
3. patients with NIHSS scores of 4 to 22 and limb weakness including motor arm or motor leg score ≥2 of NIHSS;
4. patients within 6 hours of onset or the last time known to be symptom free (within 6 hours of the start of sleep for ischemic stroke patients with onset during sleep), and who receive a CT test before the clinical study;
5. Informed consent should be signed from the patient or patient's legally authorized representative;
6. patients with premorbid mRS score of 0~1;
7. patients with no history of myocardial infarction within last 3 months;
8. patients with no heart, liver, kidney and lung function deficit;
9. patients with no hemorrhagic diseases within last 3 months;
10. patients with no haematological diseases.

Exclusion Criteria:

1. Any contraindication to CT and MRI (e.g., metal implants such as pacemakers, claustrophobia);
2. Stroke caused by posterior circulation ischemia, or transient ischemic attack (TIA);
3. Acute intracranial hemorrhage, intracranial neoplasm, cobweb hemorrhage, cerebritis or other non-acute ischemic stroke and cerebral arteriovenous malformation;
4. Endovascular treatment within 6 hours of onset, such as mechanical embolectomy, stent angioplasty or arteriovenous bridge treatment;
5. Pregnant or lactating women. Note: the pregnancy test of fertile women must be negative before randomization into groups, and female patients must take appropriate contraceptive methods at least for 3 weeks prior to the clinical study and over the next 7 days following the last injection of test drugs;
6. Pre-existing medical, neurologic, or psychiatric diseases that would confound the neurologic, functional, or imaging evaluations, such as persistent deficit from previous ischemic stroke;
7. Malignant tumor or other critical disease;
8. Patients with a history of epilepsy or undergoing seizure on onset of the ischemic stroke
9. A history of intracranial hemorrhage;
10. Patients with low blood pressure, or showing blood pressure lower than 90/60mmHg in three consecutive times after admission;
11. A history of severe injury and surgical operation within the last 3 months;
12. Consciousness disorder as defined as "NIHSS Ia score ≥2 ";
13. Complete atrioventricular block bradycardia;
14. Cardiac function rating above II level according to the New York heart association (NYHA) grade of cardiac function, history of congestive heart failure (CHF);
15. With primary liver and kidney disease, AST or ALT 2 times greater than upper normal limit, serum creatinine >2.0 mg/dL or >176.8 µmol/L;
16. International normalized ratio (INR) > 1.7 or current use of oral anticoagulants, except aspirin, clopidogrel, subcutaneous heparin or warfarin;
17. With bleeding tendency disease (such as hemophilia), partial thromboplastin time (PTT) > 3 ×the upper limit of normal;
18. A history of, or known current problems with, drug or alcohol abuse;
19. A irritability experience of the study drugs or drugs with similar chemical structures;
20. Participation in other clinical trials or studies before this study within the last 3 months;
21. Researchers consider that patients don't suit for the study.
22. Hepatitis B and C, HIV-positive patients

Imaging exclusion criteria:

1. patients with high density lesions associated with haemorrhage on CT scan after admission;
2. patients with significant lower density lesions of 1/3 middle cerebral artery on CT scan after admission;
3. patients with intracranial parenchymal tumors on CT scan after admission.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
The ratio of patients with NIHSS score of 0-1 or with reduction of NIHSS score of ≥4 than the baseline on 14 ± 2 day following the first injection. | days:14±2
  The ratio of patients with NIHSS score of 0-1 or with reduction of NIHSS score of ≥4 than the baseline on 14 ± 2 day following the first injection.

SECONDARY OUTCOMES:
Change from the baseline in NIHSS score on 14 ± 2, 30 ± 2 and 90 ± 7 days following the first injection. 1. Change from the baseline in NIHSS score on 14 ± 2, 30 ± 2 and 90 ± 7 days following the first injection. | days 14±2, 30±2 and 90±7
  Change from the baseline in NIHSS score on 14 ± 2, 30 ± 2 and 90 ± 7 days following the first injection.
Change from the baseline in mRS score on 14 ± 2, 30 ± 2 and 90 ± 7 days following the first injection. | days 14±2, 30±2 and 90±7
  Change from the baseline in mRS score on 14 ± 2, 30 ± 2 and 90 ± 7 days following the first injection.
Change from the baseline in Barthel Index (BI) score on 14 ± 2, 30 ± 2 and 90 ± 7 days following the first injection. | days 14±2, 30±2 and 90±7
  Change from the baseline in Barthel Index (BI) score on 14 ± 2, 30 ± 2 and 90 ± 7 days following the first injection.

OTHER OUTCOMES:
Exploratory Imaging Analysis for Infarct Measurement | day 6±1
  Change in infarct volume of the patient measured with MRI prior to the first injection of Neu2000KWL (baseline) and 6 ± 1 day following the first injection.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Wang, MD, Ph.D, Study Director — IRB of Beijing Tiantan Hospital, Capital Medical University
Locations (1):
- Beijing Stroke Association, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No